CLINICAL TRIAL: NCT00566852
Title: A Randomized, Phase III, Double-Blind, Placebo-Controlled Trial of Memantine for Prevention of Cognitive Dysfunction in Patients Receiving Whole-Brain Radiotherapy
Brief Title: Memantine in Preventing Side Effects in Patients Undergoing Whole-Brain Radiation Therapy for Brain Metastases From Solid Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RTOG-0614; CDR0000577872; NCI-2009-00735 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2007-12-01; First posted 2007-12-04 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-07

CONDITIONS: Cognitive/Functional Effects; Metastatic Cancer; Neurotoxicity; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: cognitive/functional effects; neurotoxicity; tumors metastatic to brain; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Neoplasm Metastasis; Neurotoxicity Syndromes; Brain Neoplasms | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WBRT+Memantine (Experimental): Whole brain radiation therapy (WBRT) and memantine
  Interventions: Drug: Memantine; Radiation: Whole brain radiation therapy
- WBRT+Placebo (Active Comparator): Whole brain radiation therapy (WBRT) and placebo
  Interventions: Other: Placebo; Radiation: Whole brain radiation therapy

INTERVENTIONS:
Drug: Memantine — Patients began taking memantine(by mouth) while receiving radiation therapy. Patients continued taking memantine for 24 weeks or until doctor thinks it is in their best interest to stop. They started with 5 mg once a day. After a week dose increased to 5 mg twice a day. At week 3, dose increased to 10 mg in the morning and 5 mg in the evening. Weeks 4-24, dose was 10 mg twice a day.
  Arms: WBRT+Memantine
Other: Placebo — Patients began taking placebo(by mouth) while receiving radiation therapy. Patients continued taking placebo for 24 weeks or until doctor thinks it is in their best interest to stop. They started with 5 mg once a day. After a week dose increased to 5 mg twice a day. At week 3, dose increased to 10 mg in the morning and 5 mg in the evening. Weeks 4-24, dose was 10 mg twice a day.
  Arms: WBRT+Placebo
Radiation: Whole brain radiation therapy — Whole brain radiation therapy (WBRT) once a day (2.5Gy), five days a week (Monday to Friday) for three weeks, for total fifteen treatments and 37.5 Gy

SUMMARY:
RATIONALE: Memantine may be able to decrease side effects caused by whole-brain radiation therapy. It is not yet known if memantine is effective in preventing side effects caused by whole-brain radiation therapy.

PURPOSE: This randomized phase III trial is studying memantine to see how well it works compared to a placebo in preventing side effects caused by whole-brain radiation therapy in patients with brain metastases from solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether the addition of memantine hydrochloride to whole-brain radiotherapy (WBRT) preserves cognitive function, specifically memory, as measured by the Hopkins Verbal Learning Test for delayed recall (HVLT-delayed recall), over that of placebo and WBRT in patients with brain metastases at 24 weeks from the start of drug treatment.

Secondary

* Determine whether the addition of memantine hydrochloride preserves cognitive function, specifically memory, as measured by the HVLT-delayed recall at 8 weeks, 16 weeks, and 12 months from the start of drug treatment.
* Determine whether the addition of memantine hydrochloride increases time to neurocognitive failure as measured by cognitive decline on a battery of tests including the HVLT for free recall, delayed recall, and delayed recognition; the Controlled Word Association Test (COWAT); the Trail Making Test Parts A and B (TMT); the Medical Outcomes Scale-Cognitive Functioning Subscale (MOS); and the Mini-Mental Status Examination (MMSE).
* Evaluate the potential benefit of memantine hydrochloride in change and overall quality of life, as measured by the Functional Assessment of Cancer Therapy-Brain (FACT-Br) subscale.
* Determine whether the addition of memantine hydrochloride increases progression-free survival.
* Determine whether the addition of memantine hydrochloride increases overall survival.
* Compare adverse events between the treatment arms according to the CTCAE v3.0 criteria.
* Collect serum, plasma, buffy coat cells, urine, and cerebrospinal fluid (CSF) for future translational research analyses.

OUTLINE: This is a multicenter study. Patients are stratified according to recursive partitioning analysis (RPA) prognostic class (class I vs class II with controlled systemic disease) and prior surgical therapy (none vs radiosurgery or surgical resection). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo whole-brain radiotherapy (WBRT) 5 days a week for 3 weeks (15 fractions). Patients also receive oral memantine hydrochloride once daily beginning on day 1 of WBRT and continuing for 24 weeks.
* Arm II: Patients undergo WBRT as in arm I. Patients also receive oral placebo once daily beginning on day 1 of WBRT and continuing for 24 weeks.

After completion of study treatment, patients are followed at 6 months, every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed diagnosis of a solid tumor malignancy within the past 5 years

  * If the original histologic proof of malignancy is > 5 years, then pathological (i.e., more recent) confirmation is required (e.g., from a systemic metastasis or brain metastasis)
* Brain metastases must be visible on contrast-enhanced MRI or a contrast enhanced CT scan (for patients unable to undergo MRI within the past 28 days)

  * Patients unable to undergo MRI imaging because of non-compatible devices are eligible, provided the contrast-enhanced CT scans are obtained and are of sufficient quality
  * Patients who had undergone radiosurgery or surgical resection and are planning adjuvant whole-brain radiotherapy do not have to have visible disease but do need a baseline MRI
* Must have stable systemic disease (i.e. no evidence of systemic disease progression within the past 3 months)
* Patients with brain metastases at initial presentation are eligible and do not need to demonstrate 3 months of stable scans

PATIENT CHARACTERISTICS:

Inclusion

* Karnofsky performance status 70-100%
* Serum creatinine ≤ 3 mg/dL and creatinine clearance ≥ 30 mL/min
* Total bilirubin ≤ 2.5 mg/dL
* Blood urea nitrogen (BUN) < 20 mg/dL
* Mini-mental status exam score ≥ 18
* Negative serum pregnancy test
* Fertile patients must practice adequate contraception

Exclusion

* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
* Pregnant or lactating women
* Prior allergic reaction to memantine hydrochloride
* Current alcohol or drug abuse
* Intractable seizures while on adequate anticonvulsant therapy (i.e., more than one seizure per month for the past 2 months)

PRIOR CONCURRENT THERAPY:

Inclusion

* At least 14 days but no more than 56 days since prior therapy for brain metastasis, including radiosurgery and surgical resection
* No systemic chemotherapy for 14 days prior, during, or for 14 days after completion of whole-brain radiotherapy (WBRT)

Exclusion

* Prior cranial radiotherapy

  * Patients may have received up to 3 prior WBRT treatments and still be registered and randomized on the protocol provided WBRT parameters meet protocol requirements
* Chronic short-acting benzodiazepine use

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2008-03; Primary Completion 2011-04 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul D. Brown, MD, Principal Investigator — Mayo Clinic; Christina A. Meyers, PhD, Study Chair — M.D. Anderson Cancer Center; Sherry Fox, RN, PhD, Study Chair — Bon Secours Cancer Institute at St. Mary's Hospital; Deepak Khuntia, MD, Study Chair — University of Wisconsin, Madison
Locations (235):
- United States (229):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Providence Cancer Center at Providence Hospital, Mobile, Alabama
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Arizona Oncology - Tucson, Tucson, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Auburn Radiation Oncology, Auburn, California
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Radiation Oncology Centers - Cameron Park, Cameron Park, California
  - Mercy Cancer Center at Mercy San Juan Medical Center, Carmichael, California
  - Enloe Cancer Center at Enloe Medical Center, Chico, California
  - Cancer Care Center at John Muir Health - Concord Campus, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Glendale Adventist Medical Center, Glendale, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - Radiation Oncology Center - Roseville, Roseville, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - Stanford Cancer Center, Stanford, California
  - Emanuel Regional Cancer Services at Emanuel Medical Center, Turlock, California
  - Solano Radiation Oncology Center, Vacaville, California
  - John Muir/Mt. Diablo Comprehensive Cancer Center, Walnut Creek, California
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - Rocky Mountain Cancer Centers - Colorado Springs, Colorado Springs, Colorado
  - Poudre Valley Radiation Oncology, Fort Collins, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Integrated Community Oncology Network at Southside Cancer Center, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Integrated Community Oncology Network, Jacksonville Beach, Florida
  - Integrated Community Oncology Network - Orange Park, Orange Park, Florida
  - Florida Institute of Research, Medicine and Surgery Cancer Center, Orlando, Florida
  - Florida Cancer Center - Palatka, Palatka, Florida
  - Flagler Cancer Center, Saint Augustine, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Northwest Community Hospital, Arlington Heights, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Saint John's Cancer Center at Saint John's Medical Center, Anderson, Indiana
  - Bloomington Hospital Regional Cancer Institute, Bloomington, Indiana
  - Radiation Oncology Associates Southwest, Fort Wayne, Indiana
  - Parkview Regional Cancer Center at Parkview Health, Fort Wayne, Indiana
  - Center for Cancer Care at Goshen General Hospital, Goshen, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - Central Indiana Cancer Centers - East, Indianapolis, Indiana
  - Community Regional Cancer Care at Community Hospital East, Indianapolis, Indiana
  - Community Regional Cancer Care at Community Hospital North, Indianapolis, Indiana
  - Cancer Center at Ball Memorial Hospital, Muncie, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Kansas City Cancer Centers - Southwest, Overland Park, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Norton Suburban Hospital, Louisville, Kentucky
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Harry and Jeanette Weinberg Cancer Institute at Franklin Square Hospital Center, Baltimore, Maryland
  - Good Samaritan Hospital of Maryland, Baltimore, Maryland
  - Central Maryland Oncology Center, Columbia, Maryland
  - Tate Cancer Center at Baltimore Washington Medical Center, Glen Burnie, Maryland
  - Cancer Institute at St. Joseph Medical Center, Towson, Maryland
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Charach Cancer Center at Huron Valley - Sinai Hospital, Commerce, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Great Lakes Cancer Institute at McLaren Regional Medical Center, Flint, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Albert Lea Cancer Center at Albert Lea Medical Center, Albert Lea, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Kansas City Cancer Centers - South, Kansas City, Missouri
  - Kansas City Cancer Centers - North, Kansas City, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Renown Institute for Cancer at Renown Regional Medical Center, Reno, Nevada
  - Payson Center for Cancer Care at Concord Hospital, Concord, New Hampshire
  - Elliot Regional Cancer Center at Elliot Hospital, Manchester, New Hampshire
  - Ocean Medical Center at Meridian Health, Brick, New Jersey
  - Cancer Institute of New Jersey at Cooper University Hospital - Camden, Camden, New Jersey
  - Trinitas Comprehensive Cancer Center at Trinitas Hospital, Elizabeth, New Jersey
  - Princeton Radiation Oncology Center, Jamesburg, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - University Medical Center at Princeton, Princeton, New Jersey
  - J. Phillip Citta Regional Cancer Center at Community Medical Center, Toms River, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - Radiation Oncology Associates, PA, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New York Oncology Hematology, PC at Albany Regional Cancer Care, Albany, New York
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Sands Cancer Center, Canandaigua, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Highland Hospital of Rochester, Rochester, New York
  - Lipson Cancer and Blood Center at Rochester General Hospital, Rochester, New York
  - University Radiation Oncology at Parkridge Hospital, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - New Hanover Radiation Oncology, PA, Wilmington, North Carolina
  - Trinity CancerCare Center, Minot, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Cleveland Clinic Cancer Center, Independence, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Cancer Care Center, Incorporated, Salem, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Precision Radiotherapy at University Pointe, West Chester, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Willamette Valley Cancer Center - Eugene, Eugene, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Dubs Cancer Center at Rogue Valley Medical Center, Medford, Oregon
  - Providence Cancer Center at PMCC, Medford, Oregon
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - UPMC Cancer Center at Beaver Medical Center, Beaver, Pennsylvania
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - UPMC Cancer Center at Jefferson Regional Medical Center, Clairton, Pennsylvania
  - Cancer Center at Clarion Hospital, Clarion, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Center - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - UPMC Cancer Center at the John P. Murtha Pavilion, Johnstown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC - Moon, Moon Township, Pennsylvania
  - UPMC Cancer Center - Natrona Heights, Natrona Heights, Pennsylvania
  - Jameson Memorial Hospital - North Campus, New Castle, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - UPMC - Shadyside, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC St. Margaret, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Passavant, Pittsburgh, Pennsylvania
  - UPMC Cancer Center - Upper St. Clair, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Cancer Center - Uniontown, Uniontown, Pennsylvania
  - Washington Hospital Cancer Center, Washington, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Texas Oncology, PA at Texas Cancer Center - Arlington South, Arlington, Texas
  - Texas Oncology, PA at Harris Center HEB, Bedford, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Texas Oncology, PA at Texas Cancer Center Dallas Southwest, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Texas Oncology, PA at Texas Cancer Center - Denton South, Denton, Texas
  - Klabzuba Cancer Center at Harris Methodist Fort Worth Hospital, Fort Worth, Texas
  - Longview Cancer Center, Longview, Texas
  - West Texas Cancer Center, Odessa, Texas
  - Cancer Care Centers of South Texas - Northeast, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Texas Oncology, PA at Texas Cancer Center - Sherman, Sherman, Texas
  - Texas Oncology, PA at Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Sentara Cancer Institute at Sentara Norfolk General Hospital, Norfolk, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Schiffler Cancer Center at Wheeling Hospital, Wheeling, West Virginia
  - Theda Care Cancer Institute, Appleton, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Community Memorial Hospital Cancer Care Center, Menomonee Falls, Wisconsin
  - Vince Lombardi Cancer Clinic at Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - All Saints Cancer Center at Wheaton Franciscan Healthcare, Racine, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - West Allis Memorial Hospital, West Allis, Wisconsin
- Canada (6):
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - McGill Cancer Centre at McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec

REFERENCES:
- [Derived] Brown PD, Pugh S, Laack NN, Wefel JS, Khuntia D, Meyers C, Choucair A, Fox S, Suh JH, Roberge D, Kavadi V, Bentzen SM, Mehta MP, Watkins-Bruner D; Radiation Therapy Oncology Group (RTOG). Memantine for the prevention of cognitive dysfunction in patients receiving whole-brain radiotherapy: a randomized, double-blind, placebo-controlled trial. Neuro Oncol. 2013 Oct;15(10):1429-37. doi: 10.1093/neuonc/not114. Epub 2013 Aug 16. PMID 23956241

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | WBRT+Memantine | WBRT+Placebo
Started | 278 | 276
Completed | 71 (Subjects with data available for analysis are considered to have completed the study.) | 78 (Subjects with data available for analysis are considered to have completed the study.)
Not Completed | 207 | 198
Not completed — Protocol Violation | 22 | 24
Not completed — Death | 95 | 78
Not completed — Withdrawal by Subject | 30 | 25
Not completed — Patient refusal | 37 | 37
Not completed — Not tested due to disability | 6 | 12
Not completed — Missing reason not specified | 1 | 2
Not completed — Missing reason not reported | 16 | 20

BASELINE CHARACTERISTICS:
Population: All randomized eligible patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | WBRT+Memantine | WBRT+Placebo | Total
Number analyzed (Participants) | 256 | 252 | 508
Age, Continuous [Median (Full Range); unit: years] | 60 [31 to 84] | 59 [29 to 86] | 59 [29 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 145 | 286
  Male | 115 | 107 | 222

OUTCOME MEASURES:

1. Primary Outcome: Change in the Hopkins Verbal Learning Test - Revised for Delayed Recall (HVLT-R-delayed Recall) at 24 Weeks
Description: The HVLT-R consists of 3 parts. Free call has a range of 0 to 36, delayed recall has a range from 0 to 12, and delayed recognition has a range of -12 to 12. Higher scores indicating better function in all 3 parts. Standardized scores are used by calculating an average standardized z score for each part of the HVLT-R. Change is calculated by subtracting baseline value from 24-week value. Imputation methods were used to determine values for all alive patients missing the 24 week assessment. This tool is being used to measure cognitive function, specifically memory.
Time Frame: Baseline and 24 weeks from the start of drug treatment
Population: All eligible patients with Hopkins Verbal Learning Test-Revised for delayed recall (HVLT-R delayed recall) at baseline and 24 weeks.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | WBRT+Memantine | WBRT+Placebo
Number analyzed (Participants) | 71 | 78
units on a scale | 0 [-1.67 to 0.59] | -0.9 [-2.22 to 0.55]
Statistical Analysis 1: Comparison: WBRT+Memantine vs WBRT+Placebo; Null hypothesis: patients on memantine will experience less decline than patients receiving placebo. Based on a one-sided Wilcoxon rank sum test with alpha=0.025, 221 patients per arm would be required to have 80% statistical power to detect a mean difference of 0.87 in the HVLT-R change scores between the two treatment arms. Assuming that 20% of patients may be ineligible, or die prior to the 24 week assessment, the target sample size for randomization was set to 536; Test type: Superiority or Other; p = 0.059, Wilcoxon (Mann-Whitney) — Significance level was 0.025

2. Secondary Outcome: Change in the Hopkins Verbal Learning Test - Revised for Delayed Recall (HVLT-R-delayed Recall) at 8, 16, and 52 Weeks
Description: The HVLT-R consists of 3 parts. Free call has a range of 0 to 36, delayed recall has a range from 0 to 12, and delayed recognition has a range of -12 to 12. Higher scores indicating better function in all 3 parts. Standardized scores are used by calculating an average standardized z score for each part of the HVLT-R. Change is calculated by subtracting baseline value from the respective later time point value. Imputation methods were used to determine values for all alive patients missing the post-baseline assessments. This tool is being used to measure cognitive function, specifically memory.
Time Frame: Baseline, 8, 16, and 52 weeks from the start of drug treatment
Population: Eligible patients with baseline and respective post-baseline measurements
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | WBRT+Memantine | WBRT+Placebo
Number analyzed (Participants) | 128 | 128
units on a scale
  8-weeks | -0.36 [-1.77 to 0.56] | -0.72 [-1.76 to 0]
  16-weeks: number analyzed (Participants) | 94 | 104
  16-weeks | 0 [-0.91 to 0.91] | 0 [-0.91 to 0.815]
  52-weeks: number analyzed (Participants) | 47 | 47
  52-weeks | 0 [-2 to 0.71] | 0 [-1.82 to 0.72]
Statistical Analysis 1: Comparison: WBRT+Memantine vs WBRT+Placebo; 8 weeks; Test type: Superiority; p = 0.0692, Wilcoxon (Mann-Whitney) — One-sided significance level of 0.025
Statistical Analysis 2: Comparison: WBRT+Memantine vs WBRT+Placebo; 16 weeks; Test type: Superiority; p = 0.4541, Wilcoxon (Mann-Whitney) — One-sided significance level of 0.025
Statistical Analysis 3: Comparison: WBRT+Memantine vs WBRT+Placebo; 52 weeks; Test type: Superiority; p = 0.3970, Wilcoxon (Mann-Whitney) — One-sided significance level of 0.025

3. Secondary Outcome: Median Time to Neurocognitive Failure
Description: Neurocognitive failure is defined as the first cognitive failure on any of the neurocognitive tests: the HVLT-R for immediate recall, delayed recognition, and delayed recall; the Controlled Oral Word Association Test (COWAT); the Trail-Making Test (TMT) Parts A and B. Cognitive failure for each test is defined as a post-treatment score that meets one of the following criteria: follow-up score is at least 2 standard deviations worse than the patient's personal baseline score or the patient's raw score change is greater than the reliable change index. The cumulative incidence approach was used to estimate the median time to neurocognitive failure to account for the competing risks of disease progression and death.
Time Frame: Baseline to 12 months from the start of drug treatment
Population: All randomized eligible patients with neurocognitive scores from baseline to 12 months from start of drug treatment.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | WBRT+Memantine | WBRT+Placebo
Number analyzed (Participants) | 256 | 252
years | 2.6 [2.4 to 3.7] | 2.3 [2.1 to 2.6]
Statistical Analysis 1: Comparison: WBRT+Memantine vs WBRT+Placebo; A one-sided log-rank test with alpha 0.025 accruing 221 patients/arm with 12 months of follow-up would ensure 98% statistical power to detect a 33% relative reduction in the monthly hazard rate with the use of memantine. Gray's test was used to test for a statistically significant difference in the distribution of neurocognitive failure times and Cox proportional hazards regression model was used to determine hazard ratios and 95% confidence intervals for the treatment difference; Test type: Superiority; p = 0.01, Gray's test; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.62 to 0.99]

4. Secondary Outcome: Change in Functional Assessment of Cancer Therapy With Brain Subscale (FACT-Br) at 24 Weeks
Description: The FACT-Br is a 50-question self-report questionnaire contains the following domains (scales): Physical well-being (7 questions), social/family well-being (7 questions), emotional well-being (6 questions), functional well-being (7 questions) and brain cancer subscale which contains concerns relevant to patients with brain tumors (23 questions). Each question has a value 0-4. For some questions a higher indicates better outcome and others are the opposite. The former are summed as is, the latter are reversed in value before adding, such that each domain ranges from 0 to 4 times the number of questions in the domain, with 0 indicating worst and the highest possible value indicating best outcome. The FACT-Br total is obtained by adding all domains together if the overall question response rate is greater than 80%. Total scores on the FACT-Br range from 0 to 184 with lower scores indicating declining quality of life. Change is calculated as baseline score subtracted from 24-week score.
Time Frame: Baseline and 24 weeks from start of treatment
Population: Eligible patients with FACT-Br score at baseline and 24 weeks.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | WBRT+Memantine | WBRT+Placebo
Number analyzed (Participants) | 71 | 66
units on a scale | 0 [-14 to 16] | 1 [-10 to 12]
Statistical Analysis 1: Comparison: WBRT+Memantine vs WBRT+Placebo; Assuming normally distributions, the two sample t-test assuming equal variances would be used to compare the arms at the 0.025 significance level. If normality assumptions were not met, the Wilcoxon rank sum would be used; Test type: Superiority; p = 0.77, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Median Progression-free Survival Time
Description: Disease progression is defined as the first of the following events: an increase of at least 50% for lesions less than or equal to 1cm, an increase of least 25% for lesions greater than 1cm, appearance of any new brain metastases. Failure for progression-free survival is disease progression or death. Median progression-free survival was estimated using the Kaplan-Meier method.
Time Frame: From randomization to date of progression, death or last follow-up. Analysis occurs at the same time as the primary outcome. Patients are followed until death and all follow-up collected at time of analysis is used.
Population: All eligible patients
Measure: Mean (Inter-Quartile Range); unit: months
Arm/Group | WBRT+Memantine | WBRT+Placebo
Number analyzed (Participants) | 256 | 252
months | 4.7 [3.7 to 5.6] | 5.5 [4.8 to 6.2]
Statistical Analysis 1: Comparison: WBRT+Memantine vs WBRT+Placebo; The stratified log-rank test was used to test for a statistically significant difference in survival distributions with a one-sided alpha of 0.025 . In addition, the Cox proportional hazards regression model was used to determine hazard ratios and 95% confidence intervals for the treatment difference; Test type: Superiority; p = 0.27, Log Rank; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.87 to 1.3]

6. Secondary Outcome: Overall Survival
Description: Failure for overall survival is death from any cause. Median survival was estimated using the Kaplan-Meier method.
Time Frame: From randomization to date of death or last follow-up. Analysis occurs at the same time as the primary outcome. Patients are followed until death and all follow-up collected at time of analysis is used.
Population: All eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | WBRT+Memantine | WBRT+Placebo
Number analyzed (Participants) | 256 | 252
months | 6.7 [5.3 to 10.2] | 7.8 [6.4 to 9.6]
Statistical Analysis 1: Comparison: WBRT+Memantine vs WBRT+Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.025, Log Rank; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.86 to 1.31]

ADVERSE EVENTS:
Description: Adverse events are reported for all eligible randomized patients with adverse event data. Subjects experiencing more than one of a given serious adverse event (SAE) are counted only once for that SAE. The same methodology was applied for non-serious adverse events.
Arm/Group | WBRT+Memantine | WBRT+Placebo
Serious Adverse Events (participants affected / at risk) | 80/251 | 67/246
Other Adverse Events (participants affected / at risk) | 160/251 | 166/246
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | WBRT+Memantine (N=251) | WBRT+Placebo (N=246)
Blood disorder (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Hemoglobin decreased (Blood and lymphatic system disorders) | 4 | 7
Arrhythmia supraventricular (Cardiac disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac pain (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0
Myocardial ischemia (Cardiac disorders) | 0 | 2
Pericardial effusion (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
External ear inflammation (Ear and labyrinth disorders) | 1 | 0
Hearing loss (Ear and labyrinth disorders) | 0 | 1
Eye disorder (Eye disorders) | 1 | 1
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 4
Colonic hemorrhage (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhea (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 1
Ileal perforation (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 9 | 6
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 10 | 9
Chest pain (General disorders) | 1 | 1
Death (General disorders) | 10 | 12
Disease progression (General disorders) | 12 | 10
Edema limbs (General disorders) | 1 | 2
Fatigue (General disorders) | 9 | 9
Fever (General disorders) | 1 | 1
General symptom (General disorders) | 2 | 0
Pain [NOS] (General disorders) | 1 | 0
Pain [other] (General disorders) | 1 | 0
Sudden death (General disorders) | 3 | 0
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 | 0
Eye infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 1 | 0
Infection [neck, with normal or Grade 1-2 ANC] (Infections and infestations) | 1 | 0
Infection [other] (Infections and infestations) | 1 | 2
Infectious colitis [with unknown ANC] (Infections and infestations) | 1 | 0
Infectious meningitis [with unknown ANC] (Infections and infestations) | 0 | 1
Peritoneal infection [with unknown ANC] (Infections and infestations) | 1 | 0
Pleural infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 1 | 0
Pneumonia [with Grade 3-4 ANC] (Infections and infestations) | 0 | 1
Pneumonia [with normal or Grade 1-2 ANC] (Infections and infestations) | 2 | 3
Pneumonia [with unknown ANC] (Infections and infestations) | 0 | 3
Urinary tract infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 1 | 1
Wound infection [with unknown ANC] (Infections and infestations) | 0 | 1
Arterial injury - Extremity-upper (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2
Alkaline phosphatase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1
Cardiac troponin I increased (Investigations) | 2 | 1
Creatinine increased (Investigations) | 0 | 1
INR increased (Investigations) | 2 | 0
Laboratory test abnormal (Investigations) | 1 | 1
Leukopenia (Investigations) | 3 | 2
Lymphopenia (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 3 | 1
Platelet count decreased (Investigations) | 1 | 3
Weight loss (Investigations) | 1 | 4
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 8 | 8
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 6 | 4
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Ataxia (Nervous system disorders) | 0 | 1
Cognitive disturbance (Nervous system disorders) | 1 | 4
Depressed level of consciousness (Nervous system disorders) | 2 | 4
Dizziness (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 6 | 1
Ischemia cerebrovascular (Nervous system disorders) | 3 | 0
Memory impairment (Nervous system disorders) | 0 | 2
Mental status changes (Nervous system disorders) | 1 | 0
Neurological disorder NOS (Nervous system disorders) | 2 | 0
Nystagmus (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 2 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 2 | 2
Speech disorder (Nervous system disorders) | 1 | 2
Syncope (Nervous system disorders) | 2 | 0
Agitation (Psychiatric disorders) | 0 | 1
Confusion (Psychiatric disorders) | 4 | 5
Depression (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Personality change (Psychiatric disorders) | 0 | 1
Psychosis (Psychiatric disorders) | 1 | 0
Bladder hemorrhage (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 | 6
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Sweating (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 1
Thrombosis (Vascular disorders) | 7 | 9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | WBRT+Memantine (N=251) | WBRT+Placebo (N=246)
Hemoglobin decreased (Blood and lymphatic system disorders) | 28 | 30
Hearing loss (Ear and labyrinth disorders) | 15 | 20
Constipation (Gastrointestinal disorders) | 34 | 25
Diarrhea (Gastrointestinal disorders) | 6 | 15
Nausea (Gastrointestinal disorders) | 56 | 67
Vomiting (Gastrointestinal disorders) | 15 | 34
Edema limbs (General disorders) | 7 | 13
Fatigue (General disorders) | 117 | 107
Dermatitis radiation (Injury, poisoning and procedural complications) | 9 | 20
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 12 | 20
Alanine aminotransferase increased (Investigations) | 11 | 17
Alkaline phosphatase increased (Investigations) | 11 | 14
Aspartate aminotransferase increased (Investigations) | 6 | 15
Laboratory test abnormal (Investigations) | 12 | 14
Leukopenia (Investigations) | 14 | 13
Lymphopenia (Investigations) | 20 | 9
Platelet count decreased (Investigations) | 18 | 15
Weight loss (Investigations) | 22 | 27
Anorexia (Metabolism and nutrition disorders) | 35 | 35
Hyperglycemia (Metabolism and nutrition disorders) | 28 | 21
Hypoalbuminemia (Metabolism and nutrition disorders) | 18 | 15
Hyponatremia (Metabolism and nutrition disorders) | 19 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 21
Muscle weakness (Musculoskeletal and connective tissue disorders) | 7 | 14
Ataxia (Nervous system disorders) | 8 | 14
Dizziness (Nervous system disorders) | 21 | 31
Headache (Nervous system disorders) | 52 | 48
Memory impairment (Nervous system disorders) | 15 | 23
Peripheral motor neuropathy (Nervous system disorders) | 14 | 13
Peripheral sensory neuropathy (Nervous system disorders) | 24 | 15
Seizure (Nervous system disorders) | 6 | 13
Taste alteration (Nervous system disorders) | 8 | 14
Depression (Psychiatric disorders) | 13 | 15
Insomnia (Psychiatric disorders) | 21 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 21
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 32 | 25
Alopecia (Skin and subcutaneous tissue disorders) | 68 | 65

LIMITATIONS AND CAVEATS:
Given the poor compliance of the HVLT-R at 24 weeks, there was only 35% statistical power to detect the hypothesized effect size. Please see linked manuscript.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.